CLINICAL TRIAL: NCT04057391
Title: Understanding Patient Experience and Preferences for the QT Scanner Compared to Mammography
Status: Suspended | Type: Observational
Why Stopped: This study was suspended by QTultrasound as other studies were reprioritized.
Sponsor: QT Ultrasound LLC (Industry)
Collaborators: Analysis Group, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: QT MG PRE Phase 1
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer Screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- QT Scanner in comparison to mammography: Women who have experience with both technologies (QT Scanner/Breast mammography
  Interventions: Diagnostic Test: QT Scanner

INTERVENTIONS:
Diagnostic Test: QT Scanner — Diagnostic test that is repeatable, non-invasive imaging tool for the early and accurate detection of breast cancer, breast abnormalities, and musculoskeletal findings. Comparing with mammography, the QT Scanner uses harmless soundwaves to screen and diagnose the breast.
  Other Names: Quantitative Transmission Ultrasound Breast Scanner-1

SUMMARY:
This study aims to characterize patient experience, satisfaction and preference for use of the QT Scanner in comparison to mammography by directly engaging women who have experience with both technologies.

DETAILED DESCRIPTION:
The objectives will be addressed by first conducting structured one-on-one interviews with about 20 women (Qualitative Phase), and then administering a web-based patient survey with quantitative measurements in about 200 women (Quantitative Phase). The current Protocol registration pertains to the first, qualitative phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Have used the QT Scanner
* Have used mammography
* Speak English
* Willing to provide consent and participate in the survey

Exclusion Criteria:

• Excluded if all Inclusion Criteria are not met

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study target population are women who have experience with both the QT Scanner and mammography.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative phase: structured one-on-one interviews | 30 days
  one-on-one interviews will be conducted by trained professionals with about 20 women

CONTACTS AND LOCATIONS:
Locations (1):
- Analysis Group, Inc., Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acquadro C, Berzon R, Dubois D, Leidy NK, Marquis P, Revicki D, Rothman M; PRO Harmonization Group. Incorporating the patient's perspective into drug development and communication: an ad hoc task force report of the Patient-Reported Outcomes (PRO) Harmonization Group meeting at the Food and Drug Administration, February 16, 2001. Value Health. 2003 Sep-Oct;6(5):522-31. doi: 10.1046/j.1524-4733.2003.65309.x. PMID 14627058
- [Background] Blumen H, Fitch K, Polkus V. Comparison of Treatment Costs for Breast Cancer, by Tumor Stage and Type of Service. Am Health Drug Benefits. 2016 Feb;9(1):23-32. PMID 27066193
- [Background] Johnson FR, Zhou M. Patient Preferences in Regulatory Benefit-Risk Assessments: A US Perspective. Value Health. 2016 Sep-Oct;19(6):741-745. doi: 10.1016/j.jval.2016.04.008. PMID 27712700
- See also: National Cancer Institute S, Epidemiology, and End Results Program,. Cancer Stat Facts: Female Breast Cancer. — https://seer.cancer.gov/statfacts/html/breast.html
- See also: National Breast Cancer Foundation I. Facts about breast cancer in the United States. 2019 — https://www.nationalbreastcancer.org/breast-cancer-facts
- See also: American Cancer Society. Breast Cancer Facts & Figures 2017-2018. — https://www.cancer.org/content/dam/cancer-org/research/cancer-facts-and-statistics/breast-cancer-facts-and-figures/breast-cancer-facts-and-figures-2017-2018.pdf